CLINICAL TRIAL: NCT01179633
Title: Acne Treatment With Active Patches Which Contains Azelaic Acid, Citric Acid,Salicylic Acid and 2% Ascorbic Acid
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oplon-Pure Science Ltd. (Industry)
Responsible Party: Dr. Avner Shemer, Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP001
Record Dates: First submitted 2010-08-05; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oplon Active Patch (Active Comparator)
  Interventions: Device: OPLON active patch
- Placebo patch (Placebo Comparator)
  Interventions: Device: Sham patch

INTERVENTIONS:
Device: OPLON active patch
  Arms: Oplon Active Patch
Device: Sham patch
  Arms: Placebo patch

SUMMARY:
The purpose of this study was to demonstrate the effect of short treatment with active OPLON patches on Acne.

DETAILED DESCRIPTION:
Patients with Acne Vulgaris were treated overnight with active patches. Effect is observed at the end of the treatment and 24 hours later.

ELIGIBILITY:
Inclusion Criteria:

* Acne Vulgaris
* Over 18 years
* Signing informed consent

Exclusion Criteria:

* Active treatment of acne
* Change in hormonal therapy
* Antibiotic treatment in a week prior to the experiment
* Sensitive skin
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Severity Score of lesion | •Severity Score of lesion [Time Frame: 24 hours following patch removal]
  Lesions were ranked by investigator according to severity whereas:
  0-clear, 1-mild, 2-moderate, 3-sever

SECONDARY OUTCOMES:
Severity Score of lesion | •Severity Score of lesion [Time Frame: 12 hours with the patch]
  0-clear, 1-mild, 2-moderate, 3-sever

CONTACTS AND LOCATIONS:
Overall Officials: Avner Shemer, MD, Principal Investigator — Laniado Medical Center
Locations (1):
- Dermatology Clinic, Netanya, Israel